CLINICAL TRIAL: NCT03091374
Title: A Proof-of-concept Study to Assess the Effect of Recombinant Human Growth Hormone on the Size of the Replication-competent Viral Reservoir in HIV-infected Individuals on Suppressive Antiretroviral Therapy
Brief Title: Impact of Recombinant Human Growth Hormone on HIV Persistence
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Collaborators: EMD Serono (Industry)
Responsible Party: Principal Investigator, Jean-Pierre Routy, Dr, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MS700149_0002
Record Dates: First submitted 2017-03-21; First posted 2017-03-27 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Human Immunodeficiency Virus; Growth Hormone Treatment
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Growth Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Growth Hormone (Experimental)
  Interventions: Drug: Somatotropin (Human)

INTERVENTIONS:
Drug: Somatotropin (Human)

SUMMARY:
Antiretroviral therapy (ART) has improved the health of more than 18 million people infected with HIV by controlling viral replication, AIDS and non-AIDS events, and by reducing the risk of transmission. However, the existence of latent viral reservoirs in long-lived memory CD4 T cells remains a hurdle to curing HIV infection; consequently patients must remain on ART for the rest of their lives. Recently, a more realistic approach under limelight is to identify strategies leading to a functional cure, which is defined as the natural control of viral reservoir by the host. Use of recombinant human growth hormone has been shown to improve immune function by several mechanisms. This study hypothesizes that treatment with recombinant human growth hormone will decrease the size of the replication competent HIV reservoir in HIV-infected immune-reconstituted individuals.

The specific study objectives include:

* To evaluate the effect of recombinant human growth hormone administration for 48 weeks on the size of the replication competent HIV reservoir
* To evaluate the safety and tolerability of recombinant human growth hormone administration for 48 weeks in HIV-infected individuals on suppressive ART.

For this purpose, the investigators will add recombinant human growth hormone treatment for the patients receiving stable ART. Approximately 22 participants will be enrolled in this study at the Chronic Viral Illness Service of the McGill University Health Centre (Montreal, Canada), which will last about 52 weeks. Participants will be treated with recombinant human growth hormone for a total of 48 weeks. The initial recombinant human growth hormone dose will be 3 mg/day (30-40 µg/kg/d) for 24 weeks administered by subcutaneous injection on an outpatient basis, followed by dose reduction to 1.5 mg/day for the final 24 weeks of the treatment period, also conducted on an outpatient basis. The study inclusion criteria include male and female participants, ≥18 and <40 years of age, with an undetectable viral load (the quantity of the HIV virus in the blood must be less than 50 copies/ml) during last 24 months and with a CD4 T-cell count ≥350 cells/mm3 obtained within 30 days prior to study entry. The findings from this study will contribute to the development of novel strategies to eradicate HIV.

DETAILED DESCRIPTION:
Antiretroviral therapy (ART) has dramatically reduced the death rate from AIDS and improved the quality of life of many HIV-infected individuals. However, ART does not eradicate HIV as demonstrated by the rapid return of viremia whenever treatment is interrupted. The possible long-term toxicity associated with ART, viral resistance, stigma and cost all contribute to the necessity of finding a cure. A sterilizing cure, in which the virus is completely eradicated, would require the elimination of all replication-competent viruses throughout the body. An alternative approach, probably more realistic, would be to aim for a kind of "cancer model" of cure, where an individual would enjoy long-term health in the absence of ART, or a disease "remission", which might be achieved after reducing the amount of residual HIV during ART (the "reservoir") to levels which the immune system can effectively control. This is commonly referred to as a functional cure in which the viral reservoir is naturally controlled by the host. Both forms of cure (sterilizing and functional) would require eliminating, or at least reducing, the reservoirs of HIV infection.

Different types of cells carry persistent HIV in virally suppressed individuals. Although myeloid cells may also contribute to HIV persistence, it is well established that the majority of replication competent viral genomes persist in memory CD4 T cells during ART. In contrast, naïve CD4 T cells are rarely infected in virally suppressed individuals. As a result of their low infection rate, the frequency of naïve cells negatively correlates with the size of the viral reservoir. Therefore, increasing the frequency of naïve cells may actively reduce the size of the latent HIV reservoir.

The thymic activity gradually decreases with age. The production of recent thymic emigrants (RTEs) is drastically reduced in the elderly, resulting in a decrease in the proportion of new naïve cells in the CD4 compartment, which is compensated by the proliferation of naïve cells in the periphery. Thus, the stability of the naïve cell pool is ensured by different mechanisms in young and elderly, with a major contribution of the thymus in young people. The study investigators preliminary data indicate that the size of the reservoir as measured by integrated DNA strongly correlates with the age of virally suppressed individuals, with younger individuals displaying a smaller reservoir). Although the mechanism underlying this remarkable association is unknown and likely to be multi-factorial, continued generation of naïve CD4 T cells during ART could lead over time to replenishment of infected memory cells with new uninfected memory cells.

Recombinant human growth hormone (rhGH) administered to ART-treated HIV infected individuals has been found to reverse thymic involution, increase total and naïve CD4 T cell counts and reduce the expression of activation and apoptosis markers. Reconstitution of the thymus in immunosuppressed adults through rhGH hormone treatment restores both HIV-specific cellular and antibody responses. Altogether, these observations suggest that the administration of rhGH may reduce the size of the latent HIV reservoir by 1) increasing the frequency of naïve cells 2) reducing the levels of immune activation and 3) restoring HIV specific immune responses, three parameters that are associated with the size of the latent HIV reservoir.

In clinical trials conducted to date using pharmacologic doses of GH, the most common adverse effects have been arthralgia and edema, both occurring in approximately 35% of patients; and myalgia, which was observed in about 30% of patients on GH. Other less common effects that are believed to be related to GH treatment include increased blood pressure, headaches, hyperglycemia and diabetes, enlargement of male breast tissue, carpal tunnel syndrome, and pancreatitis. Other, extremely rare, potential side effects that may be related to GH are allergic reactions to GH, idiopathic intracranial hypertension, hypothyroidism, and leukemia. There is conflicting evidence about whether GH increases the occurrence of lymphoma or other cancers in patients infected with HIV.

While participant enrolled in this trial might not benefit directly from the strategy, it is expected that the trial will provide useful information that relates directly to the status of the study participants (HIV infection HIV reservoirs, immunotherapeutic approaches etc.). In addition, study participants enrolled in the trial will receive compensation, clinical monitoring, laboratory monitoring and continued adherence counseling.

The investigators' primary hypothesis is that treatment with recombinant human growth hormone will result in a decrease in the size of the replication competent HIV reservoir in HIV-infected immune-reconstituted individuals. A reduction in the size of the HIV reservoir is unlikely to have any direct clinical benefits for the participants. However, this may contribute, in association with other therapies, to the development of novel strategies to eradicate HIV in the future.

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 infected male or female adults aged ≥18 and <40 years
* Able to provide written consent
* Currently on continuous ART for at least 24 months with no change in regimen in 12 weeks prior to study entry. Some modifications of ART doses during the 12 weeks prior to study entry are permitted. In addition, the change in formulation (e.g., from standard formulation to fixed-dose combination) is allowed within 12 weeks prior to study entry. A within class single drug substitution (e.g., switch from tenofovir to abacavir or raltegravir to dolutegravir) is allowed within 12 weeks prior to study entry
* CD4+ T-cell count ≥350 cells/mm3 obtained within 30 days prior to study entry.
* HIV-1 RNA level below the limit of quantification using an FDA-approved assay for at least 24 months prior to study entry and confirmed within 60 days prior to study entry. Single determinations that are between the assay quantification limit and 200 copies/mL are allowed as long as the preceding and subsequent determinations are below the level of quantification
* Female participants, may be eligible to enter and participate in the study if they are: of non-child-bearing potential (defined as physically incapable of becoming pregnant with documented tubal ligation, hysterectomy or bilateral oophorectomy), or of child- bearing potential with a negative pregnancy test at both Screening and Day 1 and agree to use one of the following methods of contraception to avoid pregnancy:

  1. Complete abstinence from penile-vaginal intercourse from 2 weeks prior to administration of IP, throughout the study, and for at least 2 weeks after discontinuation of all study medications
  2. Double barrier method (male condom/spermicide, male condom/diaphragm, diaphragm/spermicide); barrier methods must be in use at least 14 days prior to study drug administration
  3. Any intrauterine device (IUD) with published data showing that the expected failure rate is <1% per year (not all IUDs meet this criterion. IUD must be in use at least 30 days prior to first study drug administration
  4. Male partner sterilization confirmed prior to the female subject's entry into the study, and this male is the sole partner for that subject; the vasectomy must be completed 3 months prior to first study drug administration or in the alternative that a 0 sperm count will suffice
  5. Approved hormonal contraception
  6. Any other method with published data showing that the expected failure rate is <1% per year Note: Any contraception method must be used consistently, in accordance with the approved product label and for at least 2 weeks after discontinuation of recombinant human growth hormone.

Exclusion Criteria:

* Fasting glucose ≥100 mg/dL
* Hemoglobin A1c ≥ 5.7%
* ALT [serum glutamic pyruvic transaminase (SGPT)] > 2 times upper limit of normal (ULN)
* AST [serum glutamic oxaloacetic transaminase (SGOT)] > 2 x ULN
* Estimated creatinine clearance ≤ 50 mL/min by Cockcroft-Gault
* Hemoglobin < 11.5 g/dL
* Platelets <100,000/mm3
* ANC < 1000/mm3
* Any active or past history of malignancy, except for localized cutaneous Kaposi's sarcoma (fewer than 10 lesions, none of which are larger than 2 cm, and not on active therapy)
* Prior therapy with growth hormone or tesamorelin during 12 months preceding screening visit
* Unstable or untreated hypertension, defined as ≥ 160/90 mm Hg at the time of the screening visit
* History of pancreatitis, carpal tunnel syndrome (unless resolved by surgical release), diabetes mellitus, angina pectoris, coronary artery disease, or any disorder associated with moderate to severe edema (e.g. ascites, nephrotic syndrome, congestive heart failure, lymphedema)
* Acute or serious illness requiring systemic treatment and/or hospitalization within 90 days prior to study entry
* Receipt of antibiotic therapy within 30 days prior to study entry
* Chronic hepatitis C infection defined as a positive hepatitis C antibody and positive hepatitis C RNA at any time prior to study entry. Subjects who are positive for hepatitis C antibody but who are HCV RNA negative are permitted in the study
* Use of immunomodulators (e.g., interleukins, interferons, cyclosporine), HIV vaccine, systemic cytotoxic chemotherapy, or investigational therapy within 30 days prior to study entry or during study
* Known allergy/sensitivity or any hypersensitivity to components of study drug or their formulation
* Recent vaccination within 30 days prior to study entry or expected vaccination after screening but before baseline visit
* Active drug or alcohol use or dependence that, in the opinion of the site investigator, would interfere with adherence to study requirements
* Receive testosterone therapy for hypogonadism unless prior testosterone deficiency is documented
* Change in regimen or supraphysiological dose of testosterone in men (measured by elevated free testosterone above normal levels) within 2 months prior to screening
* Use of anabolic steroids, GH, GH secretagogue, GHRF products or analogs, IGF-1, or IGF binding protein 3 (IGFBP 3) within 6 months prior to screening
* Women who are lactating

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2021-03 (Actual); Study Completion 2024-12 (Actual)

PRIMARY OUTCOMES:
Change in the frequency of CD4+ T cells harbouring replication competent HIV (per 106 CD4+ T cells) between baseline (average of 2 assessments at study week -2 and 0) and 48 weeks recombinant human growth hormone administration (study week 48). | Baseline and 48 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Mcgill University Health Center, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chomont N, El-Far M, Ancuta P, Trautmann L, Procopio FA, Yassine-Diab B, Boucher G, Boulassel MR, Ghattas G, Brenchley JM, Schacker TW, Hill BJ, Douek DC, Routy JP, Haddad EK, Sekaly RP. HIV reservoir size and persistence are driven by T cell survival and homeostatic proliferation. Nat Med. 2009 Aug;15(8):893-900. doi: 10.1038/nm.1972. Epub 2009 Jun 21. PMID 19543283